CLINICAL TRIAL: NCT02777970
Title: Analgesic Efficacy of Oral Dexketoprofen Trometamol/Tramadol Hydrochloride Versus Tramadol Hydrochloride/Paracetamol: a Randomised, Double-blind, Placebo and Active-controlled, Parallel Group Study in Moderate to Severe Acute Pain After Removal of Impacted Lower Third Molar (Dexketoprofen Analgesic eVolution wIth tramaDol- DAVID Study)
Brief Title: Tramadol Hydrochloride and Dexketoprofen Trometamol for the Oral Treatment of Moderate to Severe Acute Pain Following Removal of Impacted Lower Third Molar
Acronym: DAVID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEX-TRA-06
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Acute Pain
Keywords: Acute pain; Acute moderate to severe pain; Postoperative pain; Dexketoprofen Tramadol; Dexketoprofen trometamol; Tramadol hydrochloride; Multimodal analgesia; Third molar extraction; Fixed drug combination; Paracetamol; Analgesics
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Tramadol; dexketoprofen trometamol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tramadol/Dexketoprofen (Experimental): Tramadol Hydrochloride/Dexketoprofen Trometamol 75mg/25mg film-coated tablet oral single dose;
  Placebo matching Tramadol Hydrochloride/Paracetamol 75 mg/650mg, as 2 x [37.5mg/325mg] film-coated tablets, oral single dose.
  Interventions: Drug: Tramadol Hydrochloride/Dexketoprofen Trometamol; Drug: Placebo
- Tramadol/Paracetamol (Active Comparator): Tramadol Hydrochloride/Paracetamol 75 mg/650 mg, as 2 x [37.5mg/325mg] film-coated tablets, oral single dose;
  Placebo matching Tramadol Hydrochloride/Dexketoprofen Trometamol 75mg/25mg film-coated tablet oral single dose.
  .
  Interventions: Drug: Tramadol Hydrochloride/Paracetamol; Drug: Placebo
- Placebo (Placebo Comparator): Placebo matching one film-coated tablet of Tramadol Hydrochloride/Dexketoprofen Trometamol 75mg/25mg oral single dose;
  Placebo matching two film-coated tablets of Tramadol Hydrochloride/Paracetamol 37.5mg/325mg oral single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol Hydrochloride/Dexketoprofen Trometamol
  Arms: Tramadol/Dexketoprofen
Drug: Tramadol Hydrochloride/Paracetamol
  Arms: Tramadol/Paracetamol
Drug: Placebo

SUMMARY:
The study is aimed to evaluate the analgesic efficacy of TRAM.HCl/DKP.TRIS 75mg/25mg oral fixed drug combination in comparison with TRAM.HCl /paracetamol 75mg/650mg in the treatment of moderate to severe acute pain.

DETAILED DESCRIPTION:
The present phase IV study is a randomised, double-blind, placebo and active-controlled, parallel group study in moderate to severe acute pain after removal of impacted lower third molar.

In this single-dose clinical trial patients are randomized to the following 3 treatment arms in a 2:2:1 ratio:

* TRAM.HCL/DKP.TRIS
* Paracetamol/TRAM.HCL
* Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged more than 18 years. Females participating in the study must be either non-childbearing potential or routinely using an effective method of birth control resulting in a low failure rate.
* Scheduled for outpatient surgical extraction -under local anaesthesia of lower third molar teeth, with at least one partially impacted in the mandible requiring bone manipulation.
* Pain of at least moderate intensity in the first 4 hours after the end of surgery (NRS score ≥ 4).

Exclusion Criteria:

* History of allergy or hypersensitivity to the study treatments, RM or to any other NSAIDs, opioids and acetyl salicylic acid.
* History of peptic ulcer, gastrointestinal disorders by NSAIDs or gastrointestinal bleeding or other active bleedings.
* History of any illness or condition that, in the opinion of the Investigator might pose a risk to the patient or confound the efficacy and safety results of the study.
* Patients using and not suitable for withdrawing the prohibited medications specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- Hungary (3):
  - Dr. Tóth Bagi Zoltán Fogászati Rendeloje, Budapest
  - OralMed Studio Fogászati és Szájsebészeti Kft., Budapest
  - Szegedi Tudományegyetem, Szeged
- Italy (4):
  - Ospedale Civile San Salvatore di L'Aquila, L’Aquila
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Integrata, Verona
- Poland (3):
  - Ars-Dent, Bialystok
  - Gabinet Stomatologiczny Andrzej Wojtowicz AW Clinic, Warsaw
  - Charme Clinique Klinika Stomatologii, Warsaw
- Spain (4):
  - Hospital Médico Quirúrgico de Conxo, A Coruña
  - Centro Medico Teknon, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Universidad de Valencia, Valencia
- United Kingdom (4):
  - Birmingham Community Healthcare NHS Foundation Trust, Birmingham
  - University Hospital of Wales, Cardiff
  - University of Manchester, Manchester
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gay-Escoda C, Hanna M, Montero A, Dietrich T, Milleri S, Giergiel E, Zoltan TB, Varrassi G. Tramadol/dexketoprofen (TRAM/DKP) compared with tramadol/paracetamol in moderate to severe acute pain: results of a randomised, double-blind, placebo and active-controlled, parallel group trial in the impacted third molar extraction pain model (DAVID study). BMJ Open. 2019 Feb 19;9(2):e023715. doi: 10.1136/bmjopen-2018-023715. PMID 30782886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 18 centers across 5 European countries: Hungary, Italy, Poland, Spain and the United Kingdom. The clinical phase of the study started on 28th April 2016 (first screened patient) and concluded on 14th February 2017 (last patient out).
Pre-assignment Details: A total of 792 patients were screened, of which 654 patients were randomized. One randomized patient was excluded from all the analysis populations, because of being younger than 18 years old. Prior to randomization, enrolled patients underwent a Screening period lasting up 2 weeks.
Groups:
- Tramadol/Paracetamol: Tramadol Hydrochloride/Paracetamol 75 mg/650 mg, as 2 x [37.5mg/325mg] film-coated tablets, oral single dose;
  Placebo matching Tramadol Hydrochloride/Dexketoprofen Trometamol 75mg/25mg film-coated tablet oral single dose.
Period: Overall Study
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
Started | 261 | 262 | 131
Completed | 260 | 261 | 131
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population: all patients randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo | Total
Number analyzed (Participants) | 260 | 262 | 131 | 653
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (7.48) | 27.1 (8.13) | 26.5 (7.67) | 26.9 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 104 | 53 | 309
  Male | 108 | 158 | 78 | 344
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 235 | 233 | 118 | 586
  Asian | 14 | 21 | 6 | 41
  Black or Afro-american | 7 | 3 | 6 | 16
  Other | 4 | 5 | 1 | 10
Pain Intensity at Qualification [Mean (Standard Deviation); unit: units on a scale] — Patients rate their pain intensity (PI) on e-Diary using an 11-point Numerical Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain). This PI-NRS does not include subscales.
  units on a scale | 5.0 (1.19) | 4.9 (1.12) | 4.8 (1.10) | 4.9 (1.14)

OUTCOME MEASURES:

1. Primary Outcome: TOTPAR6 (Total Pain Relief Over 6 Hours Post-dose)
Description: TOTPAR calculated as the weighted sum of the PAR scores, measured according to a 5-point VRS (Verbal Rating Scale) from 0=no relief to 4=complete relief, over 6 hours post-dose (TOTPAR6).
  The TOTPAR6 ranges from a minimum of 0 to a maximum of 24.
Time Frame: 6 hours post-dose
Population: A total of 654 patients were randomized and received the study treatments, of these one underage patient, erroneously enrolled in the study, was excluded from all the analysis populations, therefore 653 patients constituted ITT population.
Measure: Mean (Standard Deviation); unit: 5-point Verbal Rating Scale
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
Number analyzed (Participants) | 260 | 262 | 131
5-point Verbal Rating Scale | 13.0 (6.97) | 9.2 (7.65) | 1.9 (3.89)

2. Secondary Outcome: % of Patients Achieving 50% of Max TOTPAR
Description: Percentage of patients who achieved at least 50% of the maximum TOTPAR at 8 hours. In the present trial the achievable TOTPAR over 8 hours ranges between 0 and 32."
Time Frame: 8 hours post-dose
Population: ITT population
Measure: Number; unit: percentage of patients
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
Number analyzed (Participants) | 260 | 262 | 131
percentage of patients | 47.7 | 35.5 | 5.3

3. Secondary Outcome: % of Patients Achieving at Least 30% of PI (Pain Intensity) Reduction Over 8 Hours Post-dose
Description: Percentage of patients who achieve at least 30% of PI Reduction versus baseline Over 8 Hours Post-dose. Percentage change of PI is calculated using the baseline value minus the PI assessed at 8 hours post-dose divided for the baseline value, then multiplied for 100.
Time Frame: 8 hours post-dose
Population: ITT population
Measure: Number; unit: percentage of patients
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
Number analyzed (Participants) | 260 | 262 | 131
percentage of patients | 40.0 | 35.5 | 9.9

4. Secondary Outcome: Time to Confirmed FPPAR (First Perceptible Pain Relief)
Description: Time to confirmed FPPAR (time to onset of analgesia) - i.e. time to FPPAR if confirmed by experiencing Meaningful Pain Relief (MPAR)
  FPPAR and MPAR assessed by using stopwatches:
  1. 'first perceptible' PAR (FPPAR), i.e, at the moment they first felt any PAR whatsoever;
  2. 'meaningful' PAR (MPAR, ie, when the relief from pain became meaningful to them)
Time Frame: 2 hours post-dose
Population: The analysis is conducted only on active treatment arms.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol
Number analyzed (Participants) | 260 | 262
minutes | 21 [17 to 23] | 24 [20 to 27]

5. Secondary Outcome: % of Patients Requiring RM (Rescue Medication)
Description: Percentage of patients who required RM within the first over 8 hours post-dose.
Time Frame: 8 hours post-dose
Population: ITT population
Measure: Number; unit: percentage of patients
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
Number analyzed (Participants) | 260 | 262 | 131
percentage of patients | 51.2 | 55.0 | 88.5

6. Secondary Outcome: PGE (Patient Global Evaluation)
Description: PGE of the study medication (measured according to a five-point VRS from 1 = poor to 5 = excellent) at 8 hours post-dose or whenever the patient uses Rescue Medication (RM).
Time Frame: 8 hours postdose
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
Number analyzed (Participants) | 260 | 262 | 131
units on a scale | 3.6 (1.1) | 2.8 (1.4) | 1.5 (0.9)

ADVERSE EVENTS:
Time Frame: Reported treatment emergent AEs (TEAEs) include events starting after administration of study drug on or after Day 1 and on or before end of study visit Day 6+/- 1.
Description: If an AE occurs for the first time or if it worsens after study drug intake it is classified as TEAE. If a subject experienced more than 1 of a given TEAE, the subject is counted only once for that TEAE.
  Overall 654 patients received the treatment, however one patient was excluded from all the analysis populations, because of being younger than 18 years old. Thus, the safety population accounts for 653 patients.
Arm/Group | Tramadol/Dexketoprofen | Tramadol/Paracetamol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/260 | 0/262 | 0/131
Serious Adverse Events (participants affected / at risk) | 1/260 | 0/262 | 0/131
Other Adverse Events (participants affected / at risk) | 35/260 | 40/262 | 13/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol/Dexketoprofen (N=260) | Tramadol/Paracetamol (N=262) | Placebo (N=131)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol/Dexketoprofen (N=260) | Tramadol/Paracetamol (N=262) | Placebo (N=131)
Nausea (Gastrointestinal disorders) | 10 (10) | 11 (11) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 14 (14) | 0 (0)
Face oedema (General disorders) | 3 (3) | 8 (8) | 4 (4)
Dizziness (Nervous system disorders) | 6 (6) | 13 (13) | 0 (0)
Somnolence (Nervous system disorders) | 7 (7) | 4 (4) | 1 (1)
Postoperative wound infection (Infections and infestations) | 8 (8) | 2 (2) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 5 (5) | 3 (3)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT02777970/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT02777970/SAP_001.pdf